CLINICAL TRIAL: NCT00542490
Title: Phase II Trial of Vaginal Cuff Brachytherapy Followed by Carboplatin and Paclitaxel Chemotherapy in Patients With Stage I-IIb Papillary Serous, Clear Cell and Endometrioid Endometrial Cancer With High-Intermediate Risk Factors
Brief Title: Vaginal Cuff Brachytherapy Followed by Chemotherapy in Patients With Endometrioid Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1524
Record Dates: First submitted 2007-10-10; First posted 2007-10-11 (Estimated); Results first posted 2017-09-27 (Actual); Last update posted 2020-08-21 (Actual); Status verified 2020-08

CONDITIONS: Endometrial Cancer; Papillary Serous; Clear Cell Endometrial Cancer
Keywords: Endometrial cancer; Gynecologic Cancer; Vaginal Cuff Brachytherapy; Vaginal radiation
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vaginal Cuff Brachytherapy (Experimental)
  Interventions: Radiation: Vaginal Cuff Brachytherapy

INTERVENTIONS:
Radiation: Vaginal Cuff Brachytherapy — Clinical stage I-II endometrial cancer surgically staged. Stage I-II with any high-intermediate risk (H-IR) features OR Stage IIb any histology OR Stage I-II Papillary Serous or Clear Cell Histology Vaginal cuff brachytherapy Followed by Paclitaxel (175 mg/m2 over 3 hours) and carboplatin (AUC 6) Chemotherapy X 3 (high risk)

SUMMARY:
The purpose of this study is to determine the progression-free survival of patients with surgically staged, Stage I-II papillary serous, clear cell, or endometrioid carcinomas with high-intermediate risk factors treated by vaginal cuff brachytherapy followed by chemotherapy.

DETAILED DESCRIPTION:
All patients must have undergone complete surgical staging including bilateral pelvic and para-aortic lymphadenectomy. All patients will receive radiation therapy. Treatment will be delivered either by LDR or HDR brachytherapy. The treatment plan must be started at the time of enrollment. The vaginal brachytherapy should be started within 4 weeks of surgery (within 2 weeks of enrollment), in order to avoid delays in initiation of systemic therapy, which should start on post-operative day 21. The dose will be prescribed to the vaginal (mucosal) surface as defined at the surface of the applicators. Following vaginal cuff radiation therapy, all patients will receive chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have undergone specified complete surgical staging.
* Patients must be surgically staged endometrial cancer patients at high-risk for recurrence.
* Patients must have adequate bone marrow, renal and hepatic function.

Exclusion Criteria:

* Patients with recurrent disease.
* Patients with GOG performance status of 3 or 4.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2007-09; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott McMeekin, MD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vaginal Cuff Brachytherapy
Started | 23
Completed | 21
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Vaginal Cuff Brachytherapy
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 17
Age, Continuous [Mean (Full Range); unit: years] | 69 [46 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Progression-free Survival at 2 Years
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Vaginal Cuff Brachytherapy
Number analyzed (Participants) | 23
Participants | 19

2. Secondary Outcome: Number of Patients With at Least One Toxicity Related to Vaginal Cuff Brachytherapy Followed by Carboplatin and Paclitaxel Chemotherapy
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Vaginal Cuff Brachytherapy
Number analyzed (Participants) | 23
Participants | 23

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Vaginal Cuff Brachytherapy
All-Cause Mortality (participants affected / at risk) | 0/23
Serious Adverse Events (participants affected / at risk) | 1/23
Other Adverse Events (participants affected / at risk) | 1/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vaginal Cuff Brachytherapy (N=23)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Gastrointestinal bleed (Gastrointestinal disorders) | 1 (1) — gastrointestinal bleed following radiation therapy
neutropenic fever (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vaginal Cuff Brachytherapy (N=23)
Grade 4 Fatigue (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes